CLINICAL TRIAL: NCT02176161
Title: Phase II Clinical Study of Effect of Metformin on Prostate Specific Antigen Doubling Time
Brief Title: Metformin Prostate Cancer Adjuvant Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WUH 14015; 18-01662 (Other: NYU Langone Institutional Review Board)
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Results first posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer; Prostate Cancer Recurrent
Keywords: Prostate Cancer; Prostate Cancer Recurrent
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Surgery - High Risk, Undetectable prostate-specific antigen (PSA) (Experimental)
  Interventions: Drug: Metformin Hydrochloride Extended Release 750mg
- Radiation - Rising PSA (Experimental)
  Interventions: Drug: Metformin Hydrochloride Extended Release 750mg
- Surgery - Rising PSA (Experimental)
  Interventions: Drug: Metformin Hydrochloride Extended Release 750mg

INTERVENTIONS:
Drug: Metformin Hydrochloride Extended Release 750mg — Metformin Hydrochloride Extended Release 750mg twice per day for 9 months.
  Other Names: Glucophage XR; Glumetza XR

SUMMARY:
This is a Phase II clinical study to determine if Metformin can increase Prostate Specific Antigen (PSA) doubling time for patients with Prostate Cancer who have failed primary treatment with radiation, or surgical patients that are at high risk for recurrence based on surgical pathology. Men with confirmed prostate cancer and rising serum PSA levels will receive Metformin and will be monitored for PSA response and disease progression.

DETAILED DESCRIPTION:
Prostate cancer patients who have received treatment with radiation therapy or surgery, who have indicators of high-risk disease will be administered 750mg Metformin Extended Release twice per day for a period of 9 months. Metformin is an FDA-approved drug that is prescribed to treat high blood sugar levels in patients with Type 2 Diabetes. To track prostate cancer response in study participants, investigators will obtain prostate specific antigen (PSA) levels every three months for the duration of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male > 18 years of age
* Biopsy confirmed adenocarcinoma of the prostate
* Able to swallow and retain oral medication
* Hemoglobin A1C <7.0%
* Able and willing to participate in the full 12 months of the study
* Able to understand instructions related to study procedures
* Able to read and write English

Exclusion Criteria:

* Metastatic Prostate Cancer
* Prostate Specific Antigen Doubling Time < 6 months
* Prior Chemotherapy, hormonal therapy, oral glucocorticoid therapy, Gonadotropin-releasing hormone analogue therapy
* Current or previous use of 5α-reductase inhibitors, antiandrogen drugs, metformin, oral or injectable diabetes drug
* Diagnosis of Type 1 Diabetes Mellitus
* Known hypersensitivity to metformin
* any condition associated with increased risk of metformin associated lactic acidosis
* participation in any investigational or marketed drug trial within 30 days prior to screening or during study period
* any unstable, serious co-existing medical conditions including but not limited to myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to screening
* history of megaloblastic anemia
* abnormal liver function test (total bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase or serum creatinine above upper limit of normal)
* history of other malignancies, with the exception of adequately treated non-melanoma skin cancer, stage 1 melanoma, non-muscle invasive bladder cancer, or other solid tumors curatively treated with no evidence of disease for at least 5 years
* history or current evidence of substance abuse within 12 months of screening
* history of any illness (including psychiatric) that, in the opinion of the investigator, might confound the results of the study or post an additional risk to the subject

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron E Katz, MD, Principal Investigator — NYU Winthrop Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgery - High Risk, Undetectable Prostate-specific Antigen (PSA) | Radiation - Rising PSA | Surgery - Rising PSA
Started | 15 | 18 | 26
Completed | 15 | 18 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Surgery - High Risk, Undetectable Prostate-specific Antigen (PSA); Radiation - Rising PSA; Surgery - Rising PSA: Metformin Hydrochloride Extended Release 750mg twice per day for 9 months.
- Total: Total of all reporting groups
Arm/Group | Surgery - High Risk, Undetectable Prostate-specific Antigen (PSA) | Radiation - Rising PSA | Surgery - Rising PSA | Total
Number analyzed (Participants) | 15 | 18 | 26 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.02 (6.86) | 72.95 (6.86) | 72.97 (6.98) | 72.97 (6.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 15 | 18 | 26 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 9 | 11 | 17 | 37
  Unknown or Not Reported | 6 | 7 | 7 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 11 | 13 | 21 | 45
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 5 | 14
Region of Enrollment [Number; unit: participants]
  United States | 15 | 18 | 26 | 59

OUTCOME MEASURES:

1. Primary Outcome: Mean Prostate Specific Antigen (PSA) Level
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Surgery - High Risk, Undetectable Prostate-specific Antigen (PSA) | Radiation - Rising PSA | Surgery - Rising PSA
Number analyzed (Participants) | 18 | 15 | 26
ng/mL | 0.61 (0.633) | 0.70 (0.67) | 0.54 (0.66)

ADVERSE EVENTS:
Time Frame: 9 months
Description: Adverse events were monitored on a monthly basis
Arm/Group | Surgery - High Risk, Undetectable Prostate-specific Antigen (PSA) | Radiation - Rising PSA | Surgery - Rising PSA
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/15 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15 | 0/26
Other Adverse Events (participants affected / at risk) | 5/18 | 0/15 | 1/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Surgery - High Risk, Undetectable Prostate-specific Antigen (PSA) (N=18) | Radiation - Rising PSA (N=15) | Surgery - Rising PSA (N=26)
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1
Tick Bite (Infections and infestations) | 1 | 0 | 0
Left basal ganglia hemorrhage (Blood and lymphatic system disorders) | 1 | 0 | 0
right inguinal hernia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT02176161/Prot_SAP_000.pdf